CLINICAL TRIAL: NCT02111304
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Two-Part Trial to Evaluate the Efficacy, Safety, and Tolerability of iOWH032 in the Treatment of Acute Dehydrating Diarrhea in Adult and Pediatric Patients With Cholera
Brief Title: Efficacy of iOWH032 in Dehydrating Cholera
Acronym: POC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial was never initiated due to PATH executive decision.
Sponsor: PATH (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: POC Study (DDP CFT PO 202)
Record Dates: First submitted 2014-04-01; First posted 2014-04-11 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-04

CONDITIONS: Secretory Diarrhea
Keywords: cholera; diarrhea; secretory diarrhea; ORS; V. cholerae O1; iOWH032; children; pharmacokinetic; Bangladesh
MeSH Terms: conditions — Cholera; Diarrhea | interventions — IOWH-032

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part A (Adults) (Active Comparator): In Part A, approximately 170 adult patients with severe dehydrating diarrhea due to cholera will be enrolled and randomized 1:1 to receive iOWH032 500 mg or placebo TID for up to 3 days
  Interventions: Drug: iOWH032
- Part B (Pediatric) (Active Comparator): Following completion of Part A, the data and safety monitoring board (DSMB) will review the unblinded data to assess safety and efficacy and conduct a futility analysis prior to proceeding to Part B.
  Following the DSMB recommendation of dose and dosing schedule for pediatric patients, Part B will be initiated. Approximately 156 pediatric patients with severe dehydrating diarrhea due to cholera will be enrolled and randomized 1:1 to receive iOWH032 or placebo at the recommended dose and dosing regimen.
  Interventions: Drug: iOWH032

INTERVENTIONS:
Drug: iOWH032

SUMMARY:
The primary hypothesis is that administration of iOWH032 to adult and pediatric males and females with acute cholera due to V. cholerae O1 reduces stool output in the first 24 hours significantly more than does the current standard of care.

DETAILED DESCRIPTION:
This is a Phase 2, randomized, double-blind, placebo-controlled study of iOWH032 in adult patients (Part A) and then pediatric patients (Part B) with acute watery diarrhea of less than 24 hours' duration due to cholera. All subjects will be treated with standard of care (IV rehydration fluids, ORS, and azithromycin less than/equal to1 g po) in addition to study drug (iOWH032 active drug or placebo). Patients will be admitted, undergo a 4- to 6-hour screening/observation period, be randomized in the study and treated with study drug (active or placebo) for up to 3 days (ie, up to 9 doses), with a follow-up visit on Day 7.

In Part A, approximately 170 adult patients with severe dehydrating diarrhea due to cholera will be enrolled and randomized 1:1 to receive iOWH032 500 mg or placebo TID for up to 3 days. Following completion of Part A, the data and safety monitoring board (DSMB) will review the unblinded data to assess safety and efficacy and conduct a futility analysis prior to proceeding to Part B.

Following the DSMB recommendation of dose and dosing schedule for pediatric patients, Part B will be initiated. Approximately 156 pediatric patients with severe dehydrating diarrhea due to cholera will be enrolled and randomized 1:1 to receive iOWH032 or placebo at the recommended dose and dosing regimen.

The primary efficacy population for Parts A and B will consist of patients who tolerate the first 3 doses of study drug (0, 8, and 16 hours post-randomization) without vomiting and whose diagnosis is subsequently confirmed by a positive culture for V. cholerae O1.

The International Centre for Diarrhoeal Disease Research, Bangladesh (icddr,b) Ethics Committee and Western Institutional Review Board (WIRB) will be informed of any serious adverse event (SAE). Occurrence of 2 or more drug-related SAEs within a group of 10 patients (20% of cumulative completed patients in the treatment group) in Part A or Part B will result in unblinding of those patients and review by the DSMB. The study can be halted, discontinued, or amended according to the recommendations of the icddr,b DSMB.

ELIGIBILITY:
Approximately 170 adult (male and female) patients must be enrolled to ensure that 96 patients (48 active and 48 placebo) are evaluable in Part A. In Part B, approximately 156 pediatric patients will be enrolled to ensure that 120 pediatric patients (60 active and 60 placebo) are evaluable for the analysis of 24 hour stool output, the primary outcome measure.

PART A - ADULTS

***Inclusion Criteria***

A patient will be considered eligible for participation in the study if the following inclusion criteria are satisfied on admission (Day 1) to the Dhaka Hospital of icddr,b:

* Adults aged 18 years to 55 years
* Duration of illness: History of acute watery diarrhea of less than 24 hours' duration without fever or visible blood in feces
* Clinical signs and symptoms of severe dehydration (>10% loss of body weight based on rehydration weight)
* Stool RDT and/or stool DF microscopy demonstrating presence of V. cholerae
* Must have a purging rate greater than/equal to 20 mL/kg (5 mL/kg/h) during the initial 4- to 6-hour screening/observation period, and signs of clinical dehydration must be corrected
* Written informed consent for participation in the study (see Section 6.1.2 for details of the consent process)
* Negative urine pregnancy test for all female patients
* Nonpregnant and nonlactating females of childbearing potential agree to either abstain from sex or use double barrier contraception (2 contraceptive methods at a time) during the study and until 1 month after the last dose of study drug

***Exclusion Criteria***

A patient with any of the following criteria at screening for study enrollment will not qualify for the study:

* Received antidiarrheal medication (eg, loperamide, diphenoxylate) within 7 days before screening
* Abnormal ECG findings, with the exception of sinus tachycardia, premature atrial contractions, or ECG intervals within normal limits for sinus rate
* Use of drugs metabolized predominantly via CYP2C9 within 7 days before screening (see Section 5.7)
* Concomitant infection requiring antimicrobial therapy other than the study drug that may interfere with the evaluation of either the efficacy or safety of the study drug
* Patients unwilling or unable to take part in this study or refusing to sign informed consent (patients who participate on the basis of proxy consent will be re-consented at the end of the screening/observation period; those refusing consent at that time will be excluded from further study participation)
* Patients previously enrolled in this or any other investigational study within the past 30 days

PART B - PEDIATRIC

***Inclusion Criteria***

A patient will be considered eligible for participation in the study if the following inclusion criteria are satisfied on admission (Day 1) to the Clinical Research Ward (CRW) of Dhaka Hospital:

* Pediatric population aged ≥ 5 years to < 18 years of age
* Duration of illness: History of acute watery diarrhea of less than 24 hours' duration without fever or visible blood in feces
* Clinical signs and symptoms of severe dehydration (>10% loss of body weight based on rehydration weight)
* Stool RDT and/or stool DF microscopy demonstrating presence of V. cholerae
* Must have a purging rate ≥5 mL/kg/h average during the initial 4- to 6-hour screening/observation period and signs of clinical dehydration must be corrected
* Parental consent for all pediatric patients participating in the study and written informed assent for children aged 11-17 years (see Section 6.1.2 for details of the consent process)
* Negative urine pregnancy test for female postmenarchal patients
* Nonpregnant and nonlactating females of childbearing potential agree to either abstain from sex or use double-barrier contraception (2 contraceptive methods at a time) during the study and until 1 month after the last dose of study drug

***Exclusion Criteria***

A patient with any of the following criteria at screening for study enrollment will not qualify for the study:

* Received antidiarrheal medication (eg, loperamide, diphenoxylate) within 7 days before screening
* Abnormal ECG findings, with the exception of sinus tachycardia, premature atrial contractions, or ECG intervals within normal limits for sinus rate
* Use of drugs metabolized predominantly via CYP2C9 (see Section 5.7) within 7 days before screening
* Concomitant infection requiring antimicrobial therapy other than the study drug that may interfere with evaluation of either the efficacy or safety of the study drug
* Children or parents/guardians unwilling or unable to take part in this study or refusing to sign informed assent/consent; applicable patients who participate on the basis of proxy assent/consent will be re-assented at the end of the screening/observation period; those refusing assent/consent at that time will be excluded from further study participation
* Patients previously enrolled in this or any other investigational study with the past 30 days

Ages: 5 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2016-01 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Output (mL/kg of body weight) of unformed stools (composite) | First 24-hour period following randomization
  The primary objectives of the study are as follows:
  * To evaluate the efficacy of iOWH032 in adults with cholera, as measured by unformed stool output in the first 24 hours after administration (Part A)
  * To determine an effective dose and dosing regimen of iOWH032 in children with cholera (Part A)
  * To evaluate the efficacy of iOWH032 at this recommended dose and dosing regimen in children with cholera (Part B)

SECONDARY OUTCOMES:
Total stool output (mL/kg body weight) (composite) | From randomization until the resolution of diarrhea, or until 3 days (72 hours post-dose) after administration of the first dose of study drug, whichever is sooner
  * Total stool output (mL/kg body weight) from randomization until the resolution of diarrhea, or until 3 days (72 hours post-dose) after administration of the first dose of study drug, whichever is sooner
  * Time to resolution of diarrhea
  * Incidence of diarrhea resolution within 48 hours and within 72 hours from the time of administration of the first dose of study drug
  * Intake of ORS solution and plain water in mL/kg from time of randomization through the last unformed stool or until 3 days (72 hours) after administration of the first dose of study drug, whichever is sooner
  * Requirement for unscheduled IV rehydration therapy (mL/kg) after randomization
  * Sodium, potassium, chloride, cAMP, parent drug, and metabolite concentrations, all in the stool
  * Sensitivity, specificity, positive and negative predictive values, and accuracy of stool DF and RDT in the diagnosis of cholera, and the impact of antibiotic therapy on DF and RDT

OTHER OUTCOMES:
Safety | Duration of Study
  The safety and tolerability endpoints for this study are AEs, clinical laboratory values, physical examination results, vital signs, and ECG findings. All patients in Part A and B of the study who receive study drug will be included in the safety analysis.
  Acceptability of the iOWH032 dispersible tablet or suspension formulation will be evaluated in Part B of the study (pediatric patients).

CONTACTS AND LOCATIONS:
Overall Officials: Wasif A Khan, MBBS/MHS, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh; KATM Ehsanul Huq, MBBS/DTM, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

REFERENCES:
- [Background] Bardhan PK, Khan WA, Ahmed S, Salam MA, Saha D, Golman D, et al. Evaluation of safety and efficacy of a novel anti-secretory anti-diarrheal agent Crofelemer (NP-303), in combination with a single oral dose of azithromycin for the treatment of acute dehydrating diarrhea caused by Vibrio cholera cholera and other Bacterial Infections: 43rd US-Japan Cooperative Medical Science Program, Kyoto, Japan, November 21, 2008.
- [Background] Boschi-Pinto C, Lanata CF, Black RE. The global burden of childhood diarrhea. Matern Child Health. 2009;3: 225-243.
- [Background] Cystic Fibrosis Mutation Database, 2009 [online] Available at: http://www.genet.sickkids.on.ca/cftr/app
- [Background] Khan WA, Saha D, Rahman A, Salam MA, Bogaerts J, Bennish ML. Comparison of single-dose azithromycin and 12-dose, 3-day erythromycin for childhood cholera: a randomised, double-blind trial. Lancet. 2002 Nov 30;360(9347):1722-7. doi: 10.1016/S0140-6736(02)11680-1. PMID 12480424
- [Background] Muanprasat C, Sonawane ND, Salinas D, Taddei A, Galietta LJ, Verkman AS. Discovery of glycine hydrazide pore-occluding CFTR inhibitors: mechanism, structure-activity analysis, and in vivo efficacy. J Gen Physiol. 2004 Aug;124(2):125-37. doi: 10.1085/jgp.200409059. PMID 15277574
- [Background] Raghupathy P, Ramakrishna BS, Oommen SP, Ahmed MS, Priyaa G, Dziura J, Young GP, Binder HJ. Amylase-resistant starch as adjunct to oral rehydration therapy in children with diarrhea. J Pediatr Gastroenterol Nutr. 2006 Apr;42(4):362-8. doi: 10.1097/01.mpg.0000214163.83316.41. PMID 16641573
- [Background] Ram PK, Choi M, Blum LS, Wamae AW, Mintz ED, Bartlett AV. Declines in case management of diarrhoea among children less than five years old. Bull World Health Organ. 2008 Mar;86(3):E-F. doi: 10.2471/blt.07.041384. No abstract available. PMID 18368194
- [Background] Saha D, Karim MM, Khan WA, Ahmed S, Salam MA, Bennish ML. Single-dose azithromycin for the treatment of cholera in adults. N Engl J Med. 2006 Jun 8;354(23):2452-62. doi: 10.1056/NEJMoa054493. PMID 16760445
- [Background] StataCorp. POWERCAL: Stata module to perform general power and sample size calculations. http://ideas.repec.org/c/boc/bocode/s422401.html. 2013. Stata Statistical Software: Release 13. StataCorp LP, College Station, TX.
- [Background] United Nations Children's Fund (UNICEF) and World Health Organization (WHO). Diarrhoea: Why children are still dying and what can be done. 2009. New York and Geneva.
- [Background] Verkman AS, Galietta LJ. Chloride channels as drug targets. Nat Rev Drug Discov. 2009 Feb;8(2):153-71. doi: 10.1038/nrd2780. Epub 2008 Jan 19. PMID 19153558
- [Background] Victora CG, Bryce J, Fontaine O, Monasch R. Reducing deaths from diarrhoea through oral rehydration therapy. Bull World Health Organ. 2000;78(10):1246-55. PMID 11100619
- [Background] World Health Organization. The rational use of drugs in the management of acute diarrhoea in children. WHO, Geneva, 1990.
- [Background] Zhou Z, Wang X, Liu HY, Zou X, Li M, Hwang TC. The two ATP binding sites of cystic fibrosis transmembrane conductance regulator (CFTR) play distinct roles in gating kinetics and energetics. J Gen Physiol. 2006 Oct;128(4):413-22. doi: 10.1085/jgp.200609622. Epub 2006 Sep 11. PMID 16966475